CLINICAL TRIAL: NCT00997659
Title: Efficacy and Safety of Chromium as a Therapeutic Intervention for Insulin Resistance Associated With Obesity
Brief Title: Chromium's Effect on Insulin Resistance in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Dennis Mynarcik, PhD, Stony Brook University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-5689
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Insulin Resistance; Obesity
Keywords: chromium picolinate; insulin resistance; obesity
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — picolinic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chromium picolinate (Experimental)
  Interventions: Dietary Supplement: chromium picolinate

INTERVENTIONS:
Dietary Supplement: chromium picolinate — 1000 mg per day

SUMMARY:
This research is to investigate the nutritional supplement chromium picolinate. A large number of people use chromium picolinate from health food stores to improve the function of the hormone insulin. The investigators are testing how effective this supplement is and are also monitoring its safety. In patients with diabetes, chromium has been shown to increase sensitivity to the hormone insulin. Since obesity can cause insensitivity or resistance to insulin, the investigators are studying obese individuals with documented insulin resistance. The investigators would like to know if chromium is also effective in treating the insulin resistance associated with obesity.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years;
2. a BMI greater or equal to 30; AND
3. an abnormal 2 hour postprandial glucose (greater than 140 mg/dl but less than 200 mg/dl) following 75 grams of a glucose load.

Exclusion Criteria:

1. positive pregnancy test (all women must have a negative pregnancy test before beginning protocol);
2. diagnosis of cancer;
3. acute illness of any sort, however, patients may be enrolled once they are stable;
4. hemoglobin less than 11.0 g/dl or hemodynamically unstable;
5. creatinine greater than or equal to 1.5 mg/dl;
6. liver dysfunction as evidenced by elevations in transaminases 2-fold higher than upper limit of normal;
7. use of certain medications within the past month (e.g., glucocorticoids).
8. untreated hypertension (systolic BP > 150 mmHG, diastolic BP>IOO mmHG);
9. patients with diabetes mellitus;
10. hypogonadism;
11. abnormal thyroid function (serum T4 < 4 or > 12; TSH < 0.35 or > 5.5) (12) any chronic liver or kidney disease; OR
12. polycystic ovarian syndrome.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure used for sample size evaluations is the (before and after) change in the rate of glucose disposal during infusion of insulin (Rd, in mg of glucose/kg lean body mass/minute) | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University GCRC, Stony Brook, New York, United States